CLINICAL TRIAL: NCT00759213
Title: Discharge Planning Assessment of Family Needs and Concerns at the Time of Infant's Discharge in the NICU
Brief Title: Discharge Planning Assessment of Family Needs
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other)
Responsible Party: Sponsor
Other Study IDs: 27215
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Family Needs / Concerns
Keywords: Discharge planning; Family needs; Family concerns; NICU; Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Any infant with a length of stay in the NICU of at least 7 days.

SUMMARY:
It is well established within pediatric and neonatal medicine that social and traditionally "non-medical" aspects of the home environment and conditions after discharge influence neonatal health both in the acute and long-term setting. Government programs and laws exist that are designed for the provision of basic pediatric health needs. Unfortunately, deficits in obtaining those services lead to preventable poor health outcomes. Hospital social workers and discharge planners are able to identify appropriate services, while lawyers are experts in ensuring those rights and services are actually obtained and delivered.

West Side Health of CCHS has implemented a medical-legal partnership along the pathways advocated by the Medical Legal Partnership for Children as part of their clinical care services. Before implementing a similar system in the NICU, a needs assessment will be performed first.

The purpose of this study is to determine what the health care team (physicians, nurses, social workers, discharge planners, etc) through our discharge planning practice establishes as the legal needs. We will collect information which is normally collected by the health care team as a part of their usual care and assessment for discharge planning. The families will not be approached directly by study staff.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the NICU
* Length of stay > 6 days
* Discharge to home

Exclusion Criteria:

* Length of stay </= 6 days
* Discharge to another hospital

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants in the NICU
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. Locke, DO, Principal Investigator — Christiana Care Health Services
Locations (2):
- United States (2):
  - Christiana Care Health Systems, Newark, Delaware
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware